CLINICAL TRIAL: NCT01394029
Title: International Sentinel Site Surveillance of Patients With Transfusional Hemosiderosis Treated With Deferasirox in Actual Practice Setting
Brief Title: Observation of Patients With Transfusional Hemosiderosis Treatment With Deferasirox
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CICL670A2301
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Transfusional Hemosiderosis
Keywords: iron overload; iron chelation; deferasirox; observational
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- deferasirox
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox
  Other Names: ICL670

SUMMARY:
This study will observe patients with transfusional hemosiderosis treated with deferasirox in actual practice setting.

ELIGIBILITY:
Inclusion Criteria:

-Patients treated with deferasirox for transfusional hemosiderosis according to the local prescribing information.

(the patients are either beginning treatment with deferasirox at the time of enrollment in the sentinel site monitoring or are currently under treatment with deferasirox and have started the treatment under prescription up to twelve months prior to enrollment in the sentinal site monitoring.

Exclusion Criteria:

* Patients with non-transfusional hemosiderosis
* Patients treated with deferasirox in an interventional clinical trial

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with deferasirox for transfusional hemosiderosis according to the local prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Serum Creatinine and liver enzyme levels | 3 years
  Observed over 3 years for each patient
Adverse Drug Reactions | 3 years
  Observed over 3 years for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Egypt (2):
  - Novartis Investigative Site, Cairo, Cairo Governorate
  - Novartis Investigative Site, Cairo
- Novartis Investigative Site, Amman, Jordan
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
- United Kingdom (2):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, London